CLINICAL TRIAL: NCT03320070
Title: A Multicenter, Randomized, Double Blind, Placebo Controlled Exploratory Study to Assess the Efficacy and Safety of Acthar Gel in Subjects With Pulmonary Sarcoidosis
Brief Title: Acthar Gel in Participants With Pulmonary Sarcoidosis
Acronym: PULSAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MNK14344100
Record Dates: First submitted 2017-10-20; First posted 2017-10-25 (Actual); Results first posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Sarcoidosis, Pulmonary
MeSH Terms: conditions — Sarcoidosis, Pulmonary

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acthar Gel in DBT Then Acthar Gel in OLE (Experimental): Participants received Acthar Gel as a 1 milliliter (mL) injection under the skin, twice weekly, for 24 weeks in the double-blind treatment (DBT) phase. Participants, who chose to continue into the optional OLE phase, then received Acthar Gel as a 1 mL injection under the skin, twice weekly, for another 24 weeks in the optional open-label extension (OLE) phase.
  Interventions: Drug: Acthar Gel
- Placebo in DBT Then Acthar Gel in OLE (Experimental): Participants received Acthar Gel matching placebo as a 1 mL injection under the skin, twice weekly, for 24 weeks in the DBT phase. Participants, who chose to continue into the optional OLE phase, then received Acthar Gel as a 1 mL injection under the skin, twice weekly, for another 24 weeks in the optional OLE phase.
  Interventions: Drug: Acthar Gel; Drug: Placebo

INTERVENTIONS:
Drug: Acthar Gel — Acthar Gel for subcutaneous (SC) injection (80 units per 1 mL)
  Other Names: H.P. Acthar Gel; Repository Corticotropin Injection
Drug: Placebo — Placebo gel for SC injection
  Other Names: Matching Placebo
  Arms: Placebo in DBT Then Acthar Gel in OLE

SUMMARY:
The purpose of this study is to find out if Acthar Gel is safe and effective to treat pulmonary sarcoidosis.

Participants will be randomly assigned (like flipping a coin) to receive a shot under their skin of Acthar Gel or a matching placebo gel that has no drug in it. They will receive their assigned shot twice a week for 24 weeks.

All participants who complete the 24-week treatment period will be eligible to receive Acthar Gel for 24 more weeks, even if they were originally in the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Has biopsy-confirmed sarcoidosis meeting American Thoracic Society criteria ≥ 1 year at screening (Visit 1)
* Has protocol-defined symptomatic pulmonary disease
* Has been receiving a stable prednisone dose between 5 mg and 40 mg (or equivalent) for pulmonary sarcoidosis, for at least 4 weeks before screening, or a stable dose of another disease-modifying anti-sarcoidosis drug for at least 3 months before screening
* Has lung function within protocol-defined parameters

Exclusion Criteria:

* Has at least a 10% change in forced vital capacity (FVC) on spirometry between Visits 1 and 2
* Has pulmonary arterial hypertension requiring treatment
* Has been treated with antitumor necrosis factor-α antibody within the past 3 months
* Has any pulmonary condition that requires treatment, therefore impeding corticosteroid tapering

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Team Leader, Study Director — Mallinckrodt
Locations (29):
- United States (29):
  - UAB Lung Health Center, Birmingham, Alabama
  - David Geffen School of Medicine, Los Angeles, California
  - National Jewish Health, Denver, Colorado
  - University of Florida Division of Pulmonary, Critical Care, and Sleep Medicine, Gainesville, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Central Florida Pulmonary Group PA, Orlando, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Laporte County Institute For Clinical Research, Michigan City, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Howard County Center for Lung and Sleep Medicine, LLC, Columbia, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Valley Medical Group, Ridgewood, New Jersey
  - Albany Medical Center, Albany, New York
  - American Health Research Inc, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Clinical Research of Gastonia, Gastonia, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Temple Lung Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Berks Schuylkill Respiratory Specialists, Ltd, Wyomissing, Pennsylvania
  - VitaLink Research - Anderson, Anderson, South Carolina
  - Medical University of South Carolina - PPDS, Charleston, South Carolina
  - Clinical Research of Charleston, Mt. Pleasant, South Carolina
  - Clinical Research of Rock Hill, Rock Hill, South Carolina
  - VitaLink Research - Spartanburg, Spartanburg, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Texas Health Science Center at Tyler, Tyler, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mirsaeidi M, Baughman RP, Sahoo D, Tarau E. Results From a Phase 4, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of Repository Corticotropin Injection for the Treatment of Pulmonary Sarcoidosis. Pulm Ther. 2023 Jun;9(2):237-253. doi: 10.1007/s41030-023-00222-2. Epub 2023 Apr 19. PMID 37072607

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 35 investigative sites in the United States from 21 February 2018 to 15 November 2021.
Pre-assignment Details: The study consisted of 2 phases: a double-blind treatment (DBT) phase and an optional open-label extension (OLE) phase. Out of the 49 participants who completed the DBT phase, 47 participants chose to continue the treatment in the optional OLE phase.
Groups:
- Acthar Gel in DBT Then Acthar Gel in OLE: Participants received Acthar Gel as a 1 milliliter (mL) injection under the skin, twice weekly, for 24 weeks in the DBT phase. Participants, who chose to continue into the optional OLE phase, then received Acthar Gel as a 1 mL injection under the skin, twice weekly, for another 24 weeks in the OLE phase.
- Placebo in DBT Then Acthar Gel in OLE: Participants received Acthar Gel matching placebo as a 1 mL injection under the skin, twice weekly, for 24 weeks in the DBT phase. Participants, who chose to continue into the optional OLE phase, then received Acthar Gel as a 1 mL injection under the skin, twice weekly, for another 24 weeks in the OLE phase.
Period: DBT Phase (Week 1 to Week 24)
Arm/Group | Acthar Gel in DBT Then Acthar Gel in OLE | Placebo in DBT Then Acthar Gel in OLE
Started | 27 | 28
Modified Intent-to-Treat Population (mITT) (The mITT population included all randomized participants who received at least 1 dose of investigational medicinal product (IMP) and who contributed any efficacy data to the study.) | 27 | 28
Safety Population (The safety population included all randomized participants who received at least 1 dose of IMP.) | 27 | 28
Completed | 24 | 25
Not Completed | 3 | 3
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 2 | 2
Period: OLE Phase (Week 25 to Week 48)
Arm/Group | Acthar Gel in DBT Then Acthar Gel in OLE | Placebo in DBT Then Acthar Gel in OLE
Started | 22 (Only participants in this arm group who opted to receive treatment in the OLE phase started this period.) | 25
Open-label Safety Population (The open-label safety population included participants who continued into the optional OLE phase and received at least one dose of IMP during the OLE phase.) | 22 | 25
Completed | 17 | 23
Not Completed | 5 | 2
Not completed — Adverse Event | 3 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Non-compliance with Study Drug | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: The safety population included all randomized participants who received at least 1 dose of IMP.
Groups:
- Acthar Gel in DBT Then Acthar Gel in OLE: Participants received Acthar Gel as a 1 mL injection under the skin, twice weekly, for 24 weeks in the DBT phase. Participants, who chose to continue into the optional OLE phase, then received Acthar Gel as a 1 mL injection under the skin, twice weekly, for another 24 weeks in the OLE phase.
- Total: Total of all reporting groups
Arm/Group | Acthar Gel in DBT Then Acthar Gel in OLE | Placebo in DBT Then Acthar Gel in OLE | Total
Number analyzed (Participants) | 27 | 28 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (9.07) | 54.8 (11.33) | 54.2 (10.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 15 | 26
  Male | 16 | 13 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 23 | 24 | 47
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 13 | 19
  White | 21 | 15 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 27 | 28 | 55

OUTCOME MEASURES:

1. Primary Outcome: DBT: Number of Participants in Each Category of Assessment Based on Forced Vital Capacity (FVC), a Pulmonary Function Test Parameter at Week 24
Description: Forced vital capacity (FVC) is a pulmonary function test parameter that indicates the amount of air that can be forcibly exhaled from the lungs after taking the deepest breath possible. It's measured by spirometry, which is a common breathing test to check lung function. Based on the absolute change of percent predicted, FVC was evaluated to determine if the condition is:
  * Improved (+1) [≥ 5% absolute change]
  * Unchanged (0) [>- 5% to < 5% absolute change], or
  * Worse (-1) [≤ -5% absolute change]
  An additional category "Missing Assessment" indicates the participants who had a missing assessment for this outcome measure.
Time Frame: Week 24
Population: The mITT population included all randomized participants who received at least 1 dose of the IMP and who contributed any efficacy data to the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Acthar Gel in DBT Then Acthar Gel in OLE | Placebo in DBT Then Acthar Gel in OLE
Number analyzed (Participants) | 27 | 28
Participants
  Improved | 10 | 7
  Unchanged | 12 | 12
  Deteriorate | 1 | 3
  Missing Assessment | 4 | 6
Statistical Analysis 1: Comparison: Acthar Gel in DBT Then Acthar Gel in OLE vs Placebo in DBT Then Acthar Gel in OLE; Test type: Superiority; p = 0.5076, Chi-squared

2. Primary Outcome: OLE: Number of Participants in Each Category of Assessment Based on FVC, a Pulmonary Function Test Parameter at Week 48
Description: as for outcome 1
Time Frame: Week 48
Population: Open-label safety population included participants who continued into the OLE phase and received at least one dose of IMP during the OLE phase
Measure: Count of Participants; unit: Participants
Arm/Group | Acthar Gel in DBT Then Acthar Gel in OLE | Placebo in DBT Then Acthar Gel in OLE
Number analyzed (Participants) | 22 | 25
Participants
  Improved | 2 | 6
  Unchanged | 13 | 11
  Deteriorate | 1 | 3
  Missing Assessment | 6 | 5

3. Primary Outcome: DBT: Number of Participants in Each Category of Assessment Based on the Diffusing Capacity of the Lungs for Carbon Monoxide (DLCO), a Pulmonary Function Test Parameter at Week 24
Description: The diffusing capacity of the lungs for carbon monoxide (DLCO) measures the ability of the lungs to transfer gas from inhaled air to the red blood cells in the blood. Participants are asked to fully inhale a low concentration of carbon monoxide and an inert tracer gas. Based on the absolute change of percent predicted, DLCO was evaluated to determine if the condition is:
  * Improved (+1) [≥ 5% absolute change]
  * Unchanged (0) [>- 5% to < 5% absolute change],
  * Worse (-1) [≤ -5% absolute change]
  An additional category "Missing Assessment" indicates the participants who had a missing assessment for this outcome measure.
Time Frame: Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Acthar Gel in DBT Then Acthar Gel in OLE | Placebo in DBT Then Acthar Gel in OLE
Number analyzed (Participants) | 27 | 28
Participants
  Improved | 5 | 4
  Unchanged | 11 | 11
  Deteriorate | 7 | 7
  Missing Assessment | 4 | 6
Statistical Analysis 1: Comparison: Acthar Gel in DBT Then Acthar Gel in OLE vs Placebo in DBT Then Acthar Gel in OLE; Test type: Superiority; p = 1.0000, Chi-squared

4. Primary Outcome: OLE: Number of Participants in Each Category of Assessment Based on the DLCO, a Pulmonary Function Test Parameter at Week 48
Description: as for outcome 3
Time Frame: Week 48
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Acthar Gel in DBT Then Acthar Gel in OLE | Placebo in DBT Then Acthar Gel in OLE
Number analyzed (Participants) | 22 | 25
Participants
  Improved | 9 | 6
  Unchanged | 3 | 6
  Deteriorate | 4 | 8
  Missing Assessment | 6 | 5

5. Primary Outcome: DBT: Number of Participants in Each Category of Assessment Based on High Resolution Computer Tomography (HRCT) at Week 24
Description: High-resolution computer tomography (HRCT) is a type of computed tomography (CT) with specific techniques to enhance image resolution. It is used in the diagnosis of various health problems, most commonly for lung disease. These images show cross sections (slices) through the lungs. HRCT imaging was evaluated by the investigator/radiologist and the central reader to determine if the condition is improved (+1), unchanged (0), or worse (-1). An additional category "Missing Assessment" indicates the participants who had a missing assessment for this outcome measure.
Time Frame: Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Acthar Gel in DBT Then Acthar Gel in OLE | Placebo in DBT Then Acthar Gel in OLE
Number analyzed (Participants) | 27 | 28
Participants
  Improved | 2 | 1
  Unchanged | 22 | 18
  Deteriorate | 0 | 4
  Missing Assessment | 3 | 5
Statistical Analysis 1: Comparison: Acthar Gel in DBT Then Acthar Gel in OLE vs Placebo in DBT Then Acthar Gel in OLE; Test type: Superiority; p = 0.0848, Chi-squared

6. Primary Outcome: OLE: Number of Participants in Each Category of Assessment Based on HRCT at Week 48
Description: as for outcome 5
Time Frame: Week 48
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Acthar Gel in DBT Then Acthar Gel in OLE | Placebo in DBT Then Acthar Gel in OLE
Number analyzed (Participants) | 22 | 25
Participants
  Improved | 1 | 6
  Unchanged | 13 | 13
  Deteriorate | 1 | 2
  Missing Assessment | 7 | 4

7. Primary Outcome: DBT: Number of Participants in Each Category of Assessment Based on the King's Sarcoidosis Questionnaire (KSQ) (General Health), a Quality of Life Parameter at Week 24
Description: King's sarcoidosis questionnaire (KSQ) (General Health) is a 28-item questionnaire for participants to indicate the status of their sarcoidosis and treatment. Each item was answered on a 7-point scale where 1 means the participant experiences the symptom all the time and 7 means the participant does not experience the symptom at all. Higher scores indicate improvement, and a change of 4 points is considered clinically meaningful. The score on the scale was evaluated to determine if the condition is:
  * Improved (+1) based on a change of ≥ 4 points
  * Unchanged (0) based on a change of >- 4 to < 4 points
  * Worse (-1) based on a change of ≤ -4 points
  An additional category "Missing Assessment" indicates the participants who had a missing assessment for this outcome measure.
Time Frame: Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Acthar Gel in DBT Then Acthar Gel in OLE | Placebo in DBT Then Acthar Gel in OLE
Number analyzed (Participants) | 27 | 28
Participants
  Improved | 11 | 7
  Unchanged | 3 | 8
  Deteriorate | 10 | 9
  Missing Assessment | 3 | 4
Statistical Analysis 1: Comparison: Acthar Gel in DBT Then Acthar Gel in OLE vs Placebo in DBT Then Acthar Gel in OLE; Test type: Superiority; p = 0.2005, Chi-squared

8. Primary Outcome: OLE: Number of Participants in Each Category of Assessment Based on the KSQ (General Health), a Quality of Life Parameter at Week 48
Description: as for outcome 7
Time Frame: Week 48
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Acthar Gel in DBT Then Acthar Gel in OLE | Placebo in DBT Then Acthar Gel in OLE
Number analyzed (Participants) | 22 | 25
Participants
  Improved | 8 | 8
  Unchanged | 2 | 5
  Deteriorate | 6 | 9
  Missing Assessment | 6 | 3

9. Primary Outcome: DBT: Number of Participants in Each Category of Assessment Based on the Fatigue Assessment Score (FAS), a Quality of Life Parameter at Week 24
Description: The fatigue assessment score (FAS) is a 10-item checklist for participants to indicate the level of their fatigue. Each item was answered on a 5-point scale where 1 means the participant does not experience the symptom all and 5 means the participant experiences the symptom all the time. Lower scores indicate improvement (less fatigue) and a change of 4 points is considered clinically meaningful. The score on the scale was evaluated to determine if the condition is:
  * Improved (+1) based on a change of ≤ -4 points
  * Unchanged (0) based on a change of >- 4 to < 4 points
  * Worse (-1) based on a change of ≥ 4 points
  An additional category "Missing Assessment" indicates the participants who had a missing assessment for this outcome measure.
Time Frame: Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Acthar Gel in DBT Then Acthar Gel in OLE | Placebo in DBT Then Acthar Gel in OLE
Number analyzed (Participants) | 27 | 28
Participants
  Improved | 6 | 6
  Unchanged | 12 | 11
  Deteriorate | 6 | 7
  Missing Assessment | 3 | 4
Statistical Analysis 1: Comparison: Acthar Gel in DBT Then Acthar Gel in OLE vs Placebo in DBT Then Acthar Gel in OLE; Test type: Superiority; p = 0.9416, Chi-squared

10. Primary Outcome: OLE: Number of Participants in Each Category of Assessment Based on FAS, a Quality of Life Parameter at Week 48
Description: as for outcome 9
Time Frame: Week 48
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Acthar Gel in DBT Then Acthar Gel in OLE | Placebo in DBT Then Acthar Gel in OLE
Number analyzed (Participants) | 22 | 25
Participants
  Improved | 7 | 4
  Unchanged | 5 | 13
  Deteriorate | 4 | 5
  Missing Assessment | 6 | 3

11. Primary Outcome: DBT: Number of Participants in Each Category of Assessment Based on Corticosteroid Taper Score in Participants Receiving Each Dose of Prednisone at Week 24
Description: Corticosteroids are first line treatment for sarcoidosis. Concerns of corticosteroid toxicity led to efforts to taper dose sooner. Participants were clinically evaluated at each visit by investigator and categorized by their condition; dose was tapered using algorithm to take them off prednisone using incremental doses of 40,30,20,10,7.5,5,2.5,0 mg, as explained with each category below.
  * Improved: When condition improved, reduce dose by 1 level
  * Unchanged:
    1. When stable condition without toxicity: At first stable visit they continue same dose; at second stable visit, reduce dose by 1 level
    2. When stable condition with toxicity: toxicity is treated; reduce dose by 1 level
  * Deteriorate: When worsening condition, increase dose by 1 or 2 levels but not >40mg/day
  Dose tapering was done based on the participant's clinical condition.
  Category "Missing Assessment" indicates participants who had a missing assessment for this outcome measure.
Time Frame: Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Acthar Gel in DBT Then Acthar Gel in OLE | Placebo in DBT Then Acthar Gel in OLE
Number analyzed (Participants) | 27 | 28
Participants
  Improved | 17 | 21
  Unchanged | 8 | 4
  Deteriorate | 0 | 0
  Missing Assessment | 2 | 3
Statistical Analysis 1: Comparison: Acthar Gel in DBT Then Acthar Gel in OLE vs Placebo in DBT Then Acthar Gel in OLE; Test type: Superiority; p = 0.1853, Chi-squared

12. Primary Outcome: OLE: Number of Participants in Each Category of Assessment Based on Corticosteroid Taper Score in Participants Receiving Each Dose of Prednisone at Week 48
Description: as for outcome 11
Time Frame: Week 48
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Acthar Gel in DBT Then Acthar Gel in OLE | Placebo in DBT Then Acthar Gel in OLE
Number analyzed (Participants) | 22 | 25
Participants
  Improved | 15 | 19
  Unchanged | 5 | 5
  Deteriorate | 0 | 0
  Missing Assessment | 2 | 1

ADVERSE EVENTS:
Time Frame: From the signing of Informed Consent Form (ICF) to follow up visit, 4 weeks after the last dose of study drug (approximately 52 weeks for a participant)
Description: The safety population included all randomized participants who received at least 1 dose of IMP. The open-label safety population included participants who continued into the OLE phase and received at least one dose of IMP during the OLE phase. As prespecified in the protocol, Adverse Events were collected and reported separately for DBT and OLE phases.
Groups:
- DBT: Acthar Gel 80 U (1 mL): Participants received Acthar Gel as a 1 mL injection under the skin, twice weekly, for 24 weeks in the DBT phase.
- DBT: Placebo: Participants received Acthar Gel matching placebo as a 1 mL injection under the skin, twice weekly, for 24 weeks in the DBT phase.
- OLE: Acthar Gel 80 U (1 mL) [Received Acthar in DBT]: Participants who received Acthar Gel in the DBT phase and opted to continue treatment in OLE phase, received Acthar Gel as a 1 mL injection under the skin, twice weekly, for 24 weeks in the OLE phase.
- OLE: Acthar Gel 80 U (1 mL) [Received Placebo in DBT]: Participants who received Acthar Gel matching placebo in the DBT phase and opted to continue treatment in OLE phase, received Acthar Gel as a 1 mL injection under the skin, twice weekly, for 24 weeks in the OLE phase.
Arm/Group | DBT: Acthar Gel 80 U (1 mL) | DBT: Placebo | OLE: Acthar Gel 80 U (1 mL) [Received Acthar in DBT] | OLE: Acthar Gel 80 U (1 mL) [Received Placebo in DBT]
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/28 | 0/22 | 0/25
Serious Adverse Events (participants affected / at risk) | 4/27 | 3/28 | 6/22 | 0/25
Other Adverse Events (participants affected / at risk) | 22/27 | 25/28 | 14/22 | 14/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DBT: Acthar Gel 80 U (1 mL) (N=27) | DBT: Placebo (N=28) | OLE: Acthar Gel 80 U (1 mL) [Received Acthar in DBT] (N=22) | OLE: Acthar Gel 80 U (1 mL) [Received Placebo in DBT] (N=25)
Uveitis (Eye disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0
Pelvic abscess (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 0
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DBT: Acthar Gel 80 U (1 mL) (N=27) | DBT: Placebo (N=28) | OLE: Acthar Gel 80 U (1 mL) [Received Acthar in DBT] (N=22) | OLE: Acthar Gel 80 U (1 mL) [Received Placebo in DBT] (N=25)
Dry eye (Eye disorders) | 2 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 2 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 2 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 1 | 3
Nausea (Gastrointestinal disorders) | 2 | 2 | 3 | 1
Chest discomfort (General disorders) | 0 | 1 | 1 | 2
Fatigue (General disorders) | 4 | 4 | 2 | 2
Injection site bruising (General disorders) | 2 | 5 | 1 | 2
Injection site swelling (General disorders) | 2 | 0 | 0 | 0
Oedema peripheral (General disorders) | 3 | 2 | 1 | 1
Peripheral swelling (General disorders) | 2 | 0 | 0 | 0
Sarcoidosis (Immune system disorders) | 3 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 2 | 3 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 2
Oral candidiasis (Infections and infestations) | 2 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 5 | 2 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 3 | 1 | 0 | 0
C-reactive protein increased (Investigations) | 1 | 0 | 2 | 1
Weight increased (Investigations) | 2 | 1 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 6 | 1 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 8 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 1 | 1 | 0
Headache (Nervous system disorders) | 4 | 7 | 1 | 0
Depression (Psychiatric disorders) | 2 | 0 | 2 | 0
Polyuria (Renal and urinary disorders) | 2 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 2 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0
Hypertension (Vascular disorders) | 2 | 1 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-05-18): https://cdn.clinicaltrials.gov/large-docs/70/NCT03320070/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/70/NCT03320070/SAP_001.pdf